CLINICAL TRIAL: NCT06577584
Title: The Profile of People with Diabetes Followed Up in the Context of the Care Trajectory Versus the Diabetes Convention
Brief Title: Comparison of Diabetes Patients - Care Trajectory Versus Convention
Status: Not yet recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S69595
Record Dates: First submitted 2024-08-19; First posted 2024-08-29 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- The Diabetes Care trajectory: The care trajectory is designed for individuals with T2DM who are treated with Glucagon-like peptide-1 (GLP-1) analogs (injectable or oral) or require 1 to 2 insulin injections per day. It can also be initiated when blood sugar-lowering medication (pills) is no longer sufficient and the use of a GLP-1 analog or insulin is being considered. The follow-up and management is mainly being taken care of by general practioners, with minor follow-up in specialised diabetes centers.
  Interventions: Other: Follow-up in the Diabetes Care Trajectory
- The Diabetes Convention: The Diabetes Convention is intended for individuals with T2DM who require specialized care due to the complexity of their insulin treatment (multiple daily insulin injections). Specialised diabetes centers in (university) hospitals are responsible for providing comprehensive follow-up and management of these patients.
  Interventions: Other: Follow-up in the Diabetes Convention

INTERVENTIONS:
Other: Follow-up in the Diabetes Care Trajectory — Being followed-up in the Diabetes Care Trajectory in Belgium
  Groups: The Diabetes Care trajectory
Other: Follow-up in the Diabetes Convention — Being followed-up in the Diabetes Convention in Belgium
  Groups: The Diabetes Convention

SUMMARY:
In Belgium, various structures and reimbursement programs are in place for managing Type 2 Diabetes Mellitus (T2DM). The Diabetes Care Trajectory is primarily utilized for patients who require a maximum of two insulin injections per day. In contrast, patients needing multiple daily insulin injections are managed under a diabetes convention program.

The Diabetes Care Trajectory has been operational since 2009. However, unlike patients in the diabetes convention program, where the profile and quality of care are regularly audited, there is limited information available regarding the profile and outcomes of patients within the Care Trajectory. This retrospective study aims to compare the profiles, including complications and quality of care, of T2DM patients across both groups.

DETAILED DESCRIPTION:
This retrospective study will collect data from T2DM patients enrolled in either the Diabetes Care Trajectory or the diabetes convention program. The data gathered will encompass quality of care, clinical status, complications, and metabolic state.

The profiles of these patient populations will be compared cross-sectionally for each year within the study period (2009-2024). Additionally, a longitudinal analysis will be conducted to examine the evolution of these profiles over the entire study period. Data will be extracted from electronic case records maintained at participating sites across Belgium.

ELIGIBILITY:
Inclusion Criteria:

* Followed in one of the NexusHealth hospitals in Belgium: https://www.nexuzhealth.com/en/why-nexuzhealth/patients/affiliated-healthcare-institutions
* Having being diagnosed with type 2 diabetes mellitus
* Followed in the Diabetes Care Trajectory or in the Diabetes Convention (group B) in Belgium Exclusion Criteria: no specific exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: T2DM patients being followed up in the Diabetes Care Trajectory or in the Diabetes Convention (group B) in Belgium
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Yearly for the entire study period (2009 - 2024)
  Glycated haemoglobin A1c

SECONDARY OUTCOMES:
Complications of diabetes | Yearly for the entire study period (2009 - 2024)
  Number of diabetes-associated complications such as retinopathy, nephropathy and macroangiopathy.
Cholesterol profile | Yearly for the entire study period (2009 - 2024)
  Total levels of cholesterol
Insulin requirements | Yearly for the entire study period (2009 - 2024)
  The need for insulin (units) on a daily basis

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Mathieu, MD,pHD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven

IPD SHARING:
Plan to Share IPD: No